CLINICAL TRIAL: NCT06472687
Title: Efects of FIFA 11+Warm-Up Program on Agilitiy, Balance And Proprioception Parameters in The Professional Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Elif Tuğçe Çil, Asistant Prof., Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: hamed
Record Dates: First submitted 2024-06-17; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIFA 11+ training group (FTG) (Experimental): The participants recruited in the FIFA 11+ training group (FTG) and control group (CG) received different warm-up program twice a week for ten weeks. The FTG received the FIFA 11+ training program and the CG received standard warm-up protocol. All subjects received the initial participant education and training program instruction. All training protocols were continued for twice weekly. The same physiotherapist applied FIFA 11+ training protocol.
  Interventions: Other: FIFA 11+ warm-up exercise training
- control group (CG) (Active Comparator): The participants recruited in the FIFA 11+ training group (FTG) and control group (CG) received different warm-up program twice a week for ten weeks. All subjects received the initial participant education and training program instruction. All training protocols were continued for twice weekly.The same physiotherapist applied FIFA 11+ training protocol. The control group performed the usual warm-up, which only included running, static and dynamic stretching.
  Interventions: Other: warm-up exercise training

INTERVENTIONS:
Other: FIFA 11+ warm-up exercise training — FIFA 11+ warm-up training program was applied to the experimentel group. control group (CG) did their usual warm-up program.
  Arms: FIFA 11+ training group (FTG)
Other: warm-up exercise training — exercise training
  Arms: control group (CG)

SUMMARY:
This study aimed to compare the effects of the FIFA 11+ warm-up program with a traditional warm-up on agility, balance, and proprioception in professional football players aged 18-30. Forty-four players were randomly assigned to either the FIFA 11+ group, which performed the program for 10 weeks, or the control group, which continued their usual warm-up routine.

ELIGIBILITY:
Inclusion Criteria:

* being 18-30 years, individuals who currently play professional football and actively participate in training and matches,
* participants with at least two years of professional football coaching experience,
* no history of any medical conditions that would hinder their ability to perform the required exercises.

Exclusion Criteria:

* a history of musculoskeletal surgery and fractures in the lower extremities,
* a history of acute injury to the musculoskeletal structures of other lower extremity joints in the last three months, affecting joint integrity and function and causing interruption of the desired physical activity for at least one day
* having a history of balance and vestibular disorders were excluded from the study.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Agility | Baseline assesment (Begining of the warm-up program), 10th week assessment (through FIFA 11+ program is completed.)
  Agility was assessed by the Illinois T test

SECONDARY OUTCOMES:
Balance | Baseline assesment (Begining of the warm-up program), 10th week assessment (through FIFA 11+ program is completed.)
  The Y balance test is used to evaluate dynamic balance.
Proprioception | Baseline assesment (Begining of the warm-up program), 10th week assessment (through FIFA 11+ program is completed.)
  Proprioception was assessed the ability to reposition the knee at 30, 45, and 60 degrees for both the player's right and left leg.

CONTACTS AND LOCATIONS:
Locations (1):
- Elif Tuğçe, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No